CLINICAL TRIAL: NCT07220434
Title: Medial Opening Wedge High Tibial Osteotomy: A Comparative Study of Plate Fixation and Self-Adjusting HTO External Fixator Techniques
Brief Title: TO Plate Fixation vs. External Fixator Comparison (HTO Plate vs. ExFix Study)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammed Cagatay Engin (Other)
Responsible Party: Sponsor-Investigator, Muhammed Cagatay Engin, Associate Professor, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTOexfix1
Record Dates: First submitted 2025-10-22; First posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Medial Compartment Osteoarthritis; Genu Varum; Varus Deformity; High Tibial Osteotomy
MeSH Terms: conditions — Genu Varum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1: Plate Fixation (Experimental): The osteotomy will be acutely corrected intraoperatively and stabilized using a Medial High Tibial locking plate.
  Interventions: Device: Medial HTO Locking Plate
- Group 2: HTO External Fixator (Active Comparator): he osteotomy will be stabilized using a Self-Adjusting HTO External Fixator. Gradual distraction (hemicallotasis) will begin 7 days post-operatively at a rate of 1 mm per day to achieve correction.
  Interventions: Device: Self-Adjusting HTO External Fixator

INTERVENTIONS:
Device: Medial HTO Locking Plate — Medial Opening Wedge High Tibial Osteotomy.
  Arms: Group 1: Plate Fixation
Device: Self-Adjusting HTO External Fixator — Medial Opening Wedge High Tibial Osteotomy.
  Arms: Group 2: HTO External Fixator

SUMMARY:
This study aims to compare the efficacy, accuracy, and functional outcomes of two different surgical stabilization techniques for medial opening wedge high tibial osteotomy (HTO) in patients with varus deformity and medial compartment osteoarthritis. Patients will be prospectively randomized into two groups: Group 1 (Plate Fixation) will receive acute (single-stage) correction and stabilization with a medial HTO locking plate. Group 2 (HTO External Fixator) will receive stabilization using a self-adjusting HTO external fixator, followed by gradual correction (hemicallotasis/distraction) starting 7 days post-operatively. The study will evaluate radiological correction, functional improvement (using the Oxford Knee Score), and complication rates over a 12-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Varus malalignment associated with medial compartment degeneration/osteoarthritis.

Indication for Medial Opening Wedge HTO. Aged 18 years or older. Willing to participate in the study and provide written informed consent.

Exclusion Criteria:

* Advanced-stage osteoarthritis (Indication for Total Knee Arthroplasty). Previous open knee surgery on the same extremity. Inability to comply with follow-up appointments. Significant comorbidities (e.g., uncontrolled diabetes, rheumatoid arthritis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Radiological Correction (Hip-Knee-Ankle Angle - HKA) | Baseline (Preoperative), 6 Weeks, 3 Months, 6 Months, and 12 Months Postoperative.
  ssessment of the mechanical axis on full-length weight-bearing radiographs (Measured in degrees).
Change in Functional Status (Oxford Knee Score - OKS) | Baseline (Preoperative), 6 Weeks, 3 Months, 6 Months, and 12 Months Postoperative.
  Patient-reported functional score assessing pain and knee function.
Change in Pain Intensity (Visual Analogue Scale - VAS) | Baseline (Preoperative), 6 Weeks, 3 Months, 6 Months, and 12 Months Postoperative
  Patient-reported pain score from 0 (no pain) to 10 (intolerable pain).

SECONDARY OUTCOMES:
Change in Femoro-Tibial Angle (FTA) | Baseline (Preoperative) and 12 Months Postoperative.
  Change in the anatomical axis measured in degrees.
Change in Mechanical Axis Percentage (MA%) | Baseline (Preoperative) and 12 Months Postoperative.
  Change in the position of the weight-bearing line on the tibial plateau.
Change in Posterior Tibial Slope (PTE) | Baseline (Preoperative) and 12 Months Postoperative.
  Change in the tibial slope measured in degrees.
Change in Patellar Height (Insall-Salvati Index) | Baseline (Preoperative) and 12 Months Postoperative.
  Change in patellar height measured by the Insall-Salvati ratio.
Incidence of Complications | Up to 12 months postoperative.
  Incidence of adverse events including pin tract infection (especially Group 2), superficial or deep infection, non-union/delayed union, lateral cortex fracture, hardware exposure, or knee stiffness.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Department of Orthopedics and Traumatology, Erzurum, Erzurum, Turkey (Türkiye)